CLINICAL TRIAL: NCT00002243
Title: A Phase 1B Dose-Range Study to Evaluate the Safety, Pharmacokinetics, and Effects of (+)-Calanolide A on Surrogate Markers in HIV-Positive Patients With No Previous Antiretroviral Therapy
Brief Title: A Study to Evaluate the Safety and Effectiveness of a New Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI), (+)-Calanolide A, in HIV-Positive Patients Who Have Never Received Anti-HIV Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarawak MediChem Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 297A; 57CL-9802
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: HIV Infections
Keywords: Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — calanolide A

INTERVENTIONS:
Drug: Calanolide A

SUMMARY:
The purpose of this study is to test the safety and effectiveness of a new non-nucleoside reverse transcriptase inhibitor (NNRTI), (+)-calanolide A, in HIV-positive patients who have never received anti-HIV treatment.

DETAILED DESCRIPTION:
Patients are randomized into 2 cohorts, with Cohort 2 receiving a higher dosage than Cohort 1. Patients in each cohort receive either (+)-calanolide A or a placebo for 14 days, followed by a 14-day follow-up period. Following study treatment, patients may elect to receive an open-label, 6-month course of anti-HIV drugs to be selected by and administered under the care of the patient's physician.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 count of at least 250 cells/mm3.
* Have an HIV count (viral load) of at least 5,000 copies/ml.
* Are at least 18 years old.

Exclusion Criteria

You will not be eligible for this study if you:

* Have received prescription or nonprescription medications within 14 days of study entry, or if you will need to take any of these medications during the study.
* Have ever received anti-HIV medications.
* Test positive for hepatitis B.
* Have received a blood (or red blood cell) transfusion within 3 months prior to study entry.
* Have severe diarrhea.
* Have severe heart, liver, kidney, or neurological (brain and spinal cord) disease.
* Have hemophilia or another blood disorder.
* Have received certain medications or vaccines within 30 days prior to study entry.
* Have received chemotherapy or radiation within 16 days prior to study entry, or if you will need either of these during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - South Florida Bioavailability Clinic, Miami, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Cook County Hosp, Chicago, Illinois
  - Univ of Maryland Institute of Human Virology, Baltimore, Maryland
  - Boston Med Ctr / Clinical Research Office, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Anderson Clinical Research / Inc, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas / Med Branch at Galveston, Galveston, Texas